CLINICAL TRIAL: NCT05494970
Title: Accompaniment of Patients by Dental Assistants in the Evaluation of Oral Hygiene During and After Radiotherapy Treatment: a Feasibility Study.
Brief Title: Accompaniment of Patients by Dental Assistants in the Evaluation of Oral Hygiene During and After Radiotherapy Treatment.
Acronym: RadioT HBD
Status: Completed | Type: Observational
Sponsor: Institut Claudius Regaud (Other)
Collaborators: Ligue contre le cancer, France (Other)
Responsible Party: Sponsor
Other Study IDs: 22VADS03
Record Dates: First submitted 2022-08-08; First posted 2022-08-10 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: ORL Cancer
Keywords: ORL Cancer; Oral hygiene; Radiotherapy; Written information guide

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with ORL cancer for which radiotherapy treatment is required.
  Interventions: Other: Accompaniment by the dental assistant.

INTERVENTIONS:
Other: Accompaniment by the dental assistant. — Inclusion visit (before radiotherapy treatment):
  * oral hygiene education (prevention of complications related to radiotherapy) will be provided by the dental assistant.
  * a written information guide on oral hygiene will be given to the patient.
  * the questionnaire entitled "Motivation and oral hygiene behavior" will be completed by the patient.
  End of study visit (three months post-radiotherapy):
  • The "Motivation and oral hygiene behavior" and the satisfaction questionnaires will be completed by the patient.

SUMMARY:
Feasibility, prospective, monocentric study aiming to evaluate the interest of a written information guide, given and explained by the dental assistant, on the improvement of the oral hygiene of patients with ORL cancer at 3 months post-radiotherapy.

The study will be conducted on a population of 44 patients with ORL cancer requiring radiation treatment.

Each patient will be followed during 3 months post-radiotherapy (follow-up for up to 12 months post-inclusion).

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years at study entry.
2. Patient with ORL cancer requiring radiotherapy (+/- associated chemotherapy).
3. Patient with a plaque index > or = 30%.
4. Patient affiliated to a social security system in France.
5. Patient having signed informed consent prior to inclusion in the study and prior to any specific procedure for the study.

Exclusion Criteria:

1. Pregnant or lactating women.
2. Any psychological, familial, geographic or sociological condition that does not allow for compliance with the medical follow-up and/or procedures outlined in the study protocol.
3. Patient who has forfeited his/her freedom by administrative or legal award or who is under legal protection (curatorship and guardianship, protection of justice).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with ORL cancer for which radiotherapy (+/- associated chemotherapy) is indicated.
Sampling Method: Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2022-10-13 (Actual); Primary Completion 2024-01-30 (Actual); Study Completion 2024-01-30 (Actual)

PRIMARY OUTCOMES:
Rate of patients with improved oral hygiene between the inclusion visit and 3 months post-radiotherapy. | 3 months per patient
  Improvement is defined as a gross decrease of at least 30% in the plaque index between the inclusion visit and 3 months post-radiotherapy. The plaque index will be evaluated using the O'Leary method.

SECONDARY OUTCOMES:
Patient satisfaction with the oral hygiene information guide and the consultations performed by the dental assistant. | 3 months per patient
  It will be evaluated by means of a satisfaction questionnaire.
The motivation of the patients towards their oral health. | 3 months per patient
  It will be evaluated with the questionnaire "Motivation and oral hygiene behavior".

CONTACTS AND LOCATIONS:
Locations (1):
- Institut Universitaire du Cancer Toulouse - Oncopole, Toulouse, France